CLINICAL TRIAL: NCT04045145
Title: A Phase 2, Open-Label, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-74788 in Pediatric Subjects With Congenital Adrenal Hyperplasia
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-74788 (Crinecerfont) in Pediatric Participants With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-74788-CAH2008
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: CAH - Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — crinecerfont

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crinecerfont 50 milligrams (mg) Twice Daily (BID) (Experimental): Crinecerfont administered orally for 14 consecutive days.
  Interventions: Drug: Crinecerfont

INTERVENTIONS:
Drug: Crinecerfont — Crinecerfont administered orally for 14 consecutive days.
  Other Names: NBI-74788

SUMMARY:
This is a Phase 2, open-label, multiple-dose, study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NBI-74788 (crinecerfont) in pediatric participants (14 to 17 years of age) with a documented medical diagnosis of classic 21-hydroxylase deficiency congenital adrenal hyperplasia (CAH).

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general health.
2. Have a medically confirmed diagnosis of classic 21-hydroxylase deficiency CAH.
3. Be on a stable regimen of steroidal treatment for CAH that is expected to remain stable throughout the study.
4. Participants of childbearing potential must be instructed on the proper use of barrier methods of contraception and agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently from screening until the final study visit or a prespecified window after the last dose of study drug, whichever is longer.
5. Participants of childbearing potential must have a negative pregnancy test at screening and negative urine pregnancy test at baseline.
6. Have a negative urine drug (for illegal drugs) and alcohol breath test at screening and baseline.
7. Be willing and able to adhere to the study regimen and study procedures described in the protocol and informed consent/assent form, including all requirements at the study center and return for the follow-up visit.

Exclusion Criteria:

1. Have a clinically significant unstable medical condition or chronic disease, or malignancy.
2. Had a medically significant illness within 30 days of screening.
3. Have a known or suspected differential diagnosis of any of the other known forms of classic CAH.
4. Have a history that includes bilateral adrenalectomy, hypopituitarism, or other condition requiring daily therapy with orally administered glucocorticoids.
5. Are pregnant or lactating females.
6. Have a history of epilepsy or serious head injury.
7. Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
8. Have hypersensitivity to any corticotropin releasing hormone antagonists.
9. Test positive at screening for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV), or have a history of a positive result.
10. Have a recent history of alcohol or drug abuse, or current evidence of substance dependence or abuse criteria.
11. Used any anticoagulants or antiplatelet therapies within 30 days before screening.
12. Have an active bleeding disorder.
13. Used any other investigational drug within 30 days before initial screening, or plans to use an investigational drug (other than the study drug) during the study.
14. Have a blood loss ≥250 mL or donated blood within 56 days or donated plasma within 7 days before baseline.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Minneapolis, Minnesota
  - Neurocrine Clinical Site, Philadelphia, Pennsylvania
  - Neurocrine Clinical Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Newfield RS, Sarafoglou K, Fechner PY, Nokoff NJ, Auchus RJ, Vogiatzi MG, Jeha GS, Giri N, Roberts E, Sturgeon J, Chan JL, Farber RH. Crinecerfont, a CRF1 Receptor Antagonist, Lowers Adrenal Androgens in Adolescents With Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2871-2878. doi: 10.1210/clinem/dgad270. PMID 37216921

RESULTS

PARTICIPANT FLOW:
Groups:
- Crinecerfont 50 mg BID: Participants received crinecerfont 50 milligrams (mg) twice daily (BID) orally for 14 consecutive days.
Period: Overall Study
Arm/Group | Crinecerfont 50 mg BID
Started | 8
Received at Least 1 Dose of Study Drug | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Crinecerfont 50 BID: Participants received crinecerfont 50 mg BID orally for 14 consecutive days.
Arm/Group | Crinecerfont 50 BID
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  White | 7
17-hydroxyprogesterone (OHP) (Morning Window Average) [Median (Inter-Quartile Range); unit: nanograms/deciliter (ng/dL)] | 7703.74 [3344.01 to 10467.50]
17-OHP (24-Hour Average) [Median (Inter-Quartile Range); unit: ng/dL] | 2739.74 [1264.84 to 5114.45]
Androstenedione Morning Window Average) [Median (Inter-Quartile Range); unit: ng/dL] | 367.88 [207.45 to 600.73]
Adrenocorticotropic hormone (ACTH) (Morning Window Average) [Median (Inter-Quartile Range); unit: picograms/milliliter (pg/mL)] | 226.23 [37.48 to 414.73]
Testosterone (Morning Window Average) [Median (Inter-Quartile Range); unit: ng/dL] — Population: Testosterone (morning window average) is presented by female and male participants separately.
  ng/dL
    Female: number analyzed (Participants) | 5
    Female | 63.50 [30.50 to 300.50]
    Male: number analyzed (Participants) | 3
    Male | 222.00 [215.50 to 355.50]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Day 14 in Serum 17-OHP Concentrations (Morning Window Average)
Description: Percent changes in 17-OHP were assessed through the collection of samples from 0700 hours to 1000 hours (morning window) both prior to study drug administration (i.e., baseline) and after 14 days of study drug dosing. The 2 samples collected during this morning window at each visit were averaged and used to determine the percent change from baseline.
Time Frame: Baseline, Day 14
Population: Pharmacodynamic (PD) analysis set included all enrolled participants who received at least one dose of study drug and had at least one PD parameter measurement at baseline and at least one PD parameter measurement at the Day 14 visit.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Crinecerfont 50 mg: Participants received crinecerfont 50 mg BID orally for 14 consecutive days.
Arm/Group | Crinecerfont 50 mg
Number analyzed (Participants) | 8
percent change | -69.48 [-89.20 to -23.05]

2. Secondary Outcome: Percent Change From Baseline to Day 14 in Serum 17-OHP Concentrations (24-hour Period)
Description: Percent changes in 17-OHP were assessed through the collection of samples for a 24-hour period prior to study drug administration (i.e., baseline) and after 14 days of study drug dosing. The average of each participant's serial sampling values at each visit where serial sampling was performed was calculated and used to determine the percent change from baseline.
Time Frame: Baseline, Day 14
Population: PD analysis set included all enrolled participants who received at least one dose of study drug and had at least one PD parameter measurement at baseline and at least one PD parameter measurement at the Day 14 visit.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Crinecerfont 50 mg
Number analyzed (Participants) | 8
percent change | -76.0 [-82.34 to -29.74]

3. Secondary Outcome: Percent Change From Baseline to Day 14 in Adrenocorticotropic Hormone (ACTH) (Morning Window Averages)
Description: Percent changes in ACTH were assessed through the collection of samples from 0700 hours to 1000 hours (morning window) both prior to study drug administration (i.e., baseline) and after 14 days of study drug dosing. The samples collected during this morning window at each visit were averaged and used to determine the percent change from baseline.
Time Frame: Baseline, Day 14
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Crinecerfont 50 mg
Number analyzed (Participants) | 8
percent change | -57.12 [-70.08 to -28.45]

4. Secondary Outcome: Percent Change From Baseline to Day 14 in Androstenedione (Morning Window Averages)
Description: Percent changes in androstenedione were assessed through the collection of samples from 0700 hours to 1000 hours (morning window) both prior to study drug administration (i.e., baseline) and after 14 days of study drug dosing. The samples collected during this morning window at each visit were averaged and used to determine the percent change from baseline.
Time Frame: Baseline, Day 14
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Crinecerfont 50 mg
Number analyzed (Participants) | 8
percent change | -58.27 [-82.22 to -11.99]

5. Secondary Outcome: Percent Change From Baseline to Day 14 in Testosterone (Morning Window Averages)
Description: Percent change in testosterone were assessed through the collection of samples from 0700 hours to 1000 hours (morning window) both prior to study drug administration (i.e., baseline) and after 14 days of study drug dosing. The samples collected during this morning window at each visit were averaged and used to determine the percent change from baseline.
Time Frame: Baseline, Day 14
Population: PD analysis set included all enrolled participants who received at least one dose of study drug and had at least one PD parameter measurement at baseline and at least one PD parameter measurement at the Day 14 visit. The overall number of participants analyzed is based on male and female participants.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Crinecerfont 50 mg
Number analyzed (Participants) | 8
percent change
  Female: number analyzed (Participants) | 5
  Female | -76.18 [-83.53 to -28.57]
  Male: number analyzed (Participants) | 3
  Male | 1.39 [-2.67 to 49.55]

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to Day 35
Description: Safety analysis set included all participants who took at least one dose of study drug and had any postbaseline safety data.
  Treatment-emergent (after dosing) or post-treatment emergent (up to 21 days after the last dose of study drug) are reported.
Arm/Group | Crinecerfont 50 mg
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crinecerfont 50 mg (N=8)
Headache (Nervous system disorders) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Blepharospasm (Eye disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04045145/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT04045145/SAP_001.pdf